CLINICAL TRIAL: NCT03883360
Title: Effects of Cannabidiol on Psychiatric Symptoms, Cognition, and Cannabis Consumption in Cannabis Users With Recent-Onset Psychosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: not funded
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Sheppard Pratt Health System (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Britta Hahn, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00082213
Record Dates: First submitted 2019-03-14; First posted 2019-03-20 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Schizophrenia Spectrum Disorders; Cannabis Use
Keywords: schizophrenia; cannabis; cannabidiol; psychosis
MeSH Terms: conditions — Schizophrenia; Marijuana Abuse; Psychotic Disorders | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to either the cannabidiol group or the placebo group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A matched placebo is employed. Only the biostatistician performing the randomization and the pharmacists will know the treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (CBD) (Experimental): Participants receive CBD daily for 12 weeks.
  Interventions: Drug: Cannabidiol (CBD)
- Placebo (Placebo Comparator): Participants receive vehicle not containing any drug daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol (CBD) — Participants receive a single dose of CBD (600 mg p.o.) per day for 12 weeks.
  Arms: Cannabidiol (CBD)
Drug: Placebo — Participants receive a single daily dose of the oil vehicle used to dissolve CBD but without any active ingredient, in the same amount as the CBD group, for 12 weeks.
  Arms: Placebo

SUMMARY:
A large proportion of people with a schizophrenia-spectrum disorder, especially in the early stages of the disease, regularly consume cannabis. Cannabis use is associated with poor prognostic outcome; however, there are no effective interventions targeted at reducing cannabis use or its deleterious effects in this population. The present trial is designed to test whether cannabidiol (CBD), a cannabinoid whose effects are in many ways antagonistic to those of Δ9-tetrahydrocannabinol (THC), can reduce psychiatric symptoms, cognitive deficits, and cannabis use in people with recent-onset psychosis who regularly consume cannabis.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled trial, evaluating the effects of a 12-week treatment course with CBD on psychiatric symptoms, cognition, and cannabis consumption in regular cannabis users with recent-onset psychosis. The study will be conducted at the Maryland Psychiatric Research Center (University of Maryland School of Medicine) and associated Early Intervention Programs in Baltimore, at the Sheppard Pratt Health System in Baltimore, and at the Psychosis Clinic of the University of California Los Angeles.

The daily dose of CBD is 600 mg (p.o.), administered as adjunct medication. Any non-exclusionary antipsychotic, antidepressant, anxiolytic, or other medication prescribed prior to the trial will be continued. Participants may, but do not have to be taking conventional antipsychotic medication.

The study will include 84 regular cannabis users with a schizophrenia-spectrum disorder who experienced their first psychotic episode within the last 5 years (90). Participants will be randomized 1:1 to either the CBD or the placebo group.

Outcome measures include psychiatric symptoms, cognition, global functioning, and drug use, and will be assessed at baseline, and every 3 or 6 weeks thereafter (depending on the measure), until the end of treatment at 12 weeks. Outcome will be assessed again at a 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, and other specified or unspecified schizophrenia spectrum and other psychotic disorder.
* Experienced a first psychotic episode within the last 5 years.
* Self-reported cannabis use at least twice/week for at least the last 4 weeks.
* THCCOOH serum levels of ≥ 5 ng/mL.
* Total score ≥45 on the 18-item version of the Brief Psychiatric Rating Scale.
* Able to give written informed consent.
* Normal or corrected to normal vision.
* If medicated, no change in psychiatric medication within the preceding 4 weeks, with no foreseeable changes.

Exclusion Criteria:

* DSM-5 diagnosis of Substance Use Disorder other that cannabis or nicotine within the last year (recreational use is not exclusionary).
* Currently undergoing active treatment for Cannabis Use Disorder other than low-level (once/week or less) psychosocial intervention.
* Uncontrolled hypertension (resting systolic BP above 150 or diastolic above 95 mm Hg).
* Cardiovascular disease, such as history of myocardial infarction and ischemia, heart failure, angina, severe arrhythmias, or EKG abnormalities (Wolf-Parkinson-White syndrome, Complete left bundle branch block, PR interval <120 ms or >200 ms, Prolonged QT interval (corrected) >500 ms, Cardiac arrhythmias as defined by PACs >3 per min or PVCs >1 per min).
* History of or current neurological illness, such as stroke, seizure disorders, neurodegenerative diseases, or organic brain syndrome.
* Intellectual disability.
* Pregnant or lactating.
* Diabetes.
* Significant kidney or liver impairment.
* Any chronic or severe infectious disease, including HIV and hepatitis.
* Cancer.
* Use of any barbiturates, diazepam, diltiazem, verapamil, protease inhibitors, any anticonvulsant medications (including valproate/valproic acid, lamotrigine, carbamazepine, and clobazam), glipizide, glyburide, warfarin, and cyclophosphamide/ ifosfamide, due to potential interaction with CBD at the metabolic level.
* Suicidal ideation currently or within last 6 months (score of >/= 3 on the Columbia Suicide Severity Rating Scale).
* Less than the lower limit of normal hemoglobin and hematocrit at screening.
* Elevated transaminase levels >3 times the ULN, accompanied by elevations in bilirubin >2 times the ULN.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2050-01 (Estimated); Primary Completion 2050-02 (Estimated); Study Completion 2050-03 (Estimated)

PRIMARY OUTCOMES:
Change in Brief Psychiatric Rating Scale (BPRS) total score | Baseline and 12 weeks
  The BPRS consists of 18 items assessing a broad range of psychiatric symptoms, including positive, negative, and affective symptoms. Each item is scored 1-7. Total scores are the sum of all items and range from 18 to 126, with larger values reflecting worse symptoms. The BPRS total score has been used widely in clinical studies of psychosis and has demonstrated reliability in assessing psychopathology across diverse psychosis populations.
Change in MATRICS Consensus Cognitive Battery (MCCB) composite score | Baseline and 12 weeks
  The MCCB is an FDA-approved assessment tool for trials of cognition-enhancing treatments in people with schizophrenia. The MCCB is comprised of the following domains: 1) Speed of Processing; 2) Attention/Vigilance; 3) Working Memory; 4) Verbal Learning; 5) Visual Learning; 6) Reasoning and Problem Solving; and 7) Social Cognition. The composite score is standardized to a T-scale (mean=50, standard deviation=10) based on healthy control normative data. Higher scores reflect better performance.
Change in Serum concentrations of THCCOOH | Baseline and 12 weeks
  THCCOOH is a THC metabolite and is used to quantify cannabis consumption. It has a long half-life (5-6 days) and thus provides a summary index of cannabis use within the last 1-2 weeks.

SECONDARY OUTCOMES:
Change in BPRS positive symptoms | Baseline and 12 weeks
  The average of four BPRS key positive symptom items (conceptual disorganization, suspiciousness, unusual thought content, and hallucinatory behavior) will be analyzed as an index of antipsychotic effects of CBD. Possible values range from 1 to 7, with larger values reflecting more severe positive symptoms.
Change in BPRS "Anxiety/Depression" subscale | Baseline and 12 weeks
  This subscale will be analyzed separately to obtain an index of the anxiolytic effects of CBD. Possible values range from 1 to 7, with larger values reflecting more anxiety/depression.
Change in State-Trait Anxiety Inventory (STAI) - State version | Baseline and 12 weeks
  The STAI-State provides another probe for potential anxiolytic effects of CBD. The participant rates 20 items about how they feel right now and a scale from 1 (not at all) to 4 (very much so). The total score is derived by adding all values and ranges from 20 to 80, with larger values indicating greater anxiety.
Change in MCCB Processing Speed subscale | Baseline and 12 weeks
  The score is standardized to a T-scale (mean=50, standard deviation=10) based on healthy control normative data. Higher scores reflect better performance.
Change in MCCB Attention/Vigilance subscale | Baseline and 12 weeks
  The score is standardized to a T-scale (mean=50, standard deviation=10) based on healthy control normative data. Higher scores reflect better performance.
Change in MCCB Working Memory subscale | Baseline and 12 weeks
  The score is standardized to a T-scale (mean=50, standard deviation=10) based on healthy control normative data. Higher scores reflect better performance.
Change in MCCB Verbal Learning subscale | Baseline and 12 weeks
  The score is standardized to a T-scale (mean=50, standard deviation=10) based on healthy control normative data. Higher scores reflect better performance.
Change in MCCB Visual Learning subscale | Baseline and 12 weeks
  The score is standardized to a T-scale (mean=50, standard deviation=10) based on healthy control normative data. Higher scores reflect better performance.
Change in MCCB Reasoning/Problem solving subscale | Baseline and 12 weeks
  The score is standardized to a T-scale (mean=50, standard deviation=10) based on healthy control normative data. Higher scores reflect better performance.
Change in MCCB Social Cognition subscale | Baseline and 12 weeks
  The score is standardized to a T-scale (mean=50, standard deviation=10) based on healthy control normative data. Higher scores reflect better performance.
Change in The UCSD Performance-Based Skills Assessment (UPSA) | Baseline and 12 weeks
  Measures ability to perform real-life tasks by standardized role-play. Scores reflect percent correct, i.e. range from 0-100, with larger scores reflecting better performance.
Change in Serum concentrations of THC | Baseline and 12 weeks
  Index of recent cannabis use.
Change in Self-reported days of cannabis use | Baseline and 12 weeks
  The reference period is the last three weeks. Thus, possible values range from 0 to 21.
Change in Cannabis Use Disorders Identification Test-Revised (CUDIT-R) | Baseline and 12 weeks
  The CUDIT-R is an 8-item questionnaire probing cannabis use frequency, amount, loss of control, and adverse consequences in the last 6 months. Each item is rated on a scale from 0 to 4. The total score is derived by summing all answers and ranges from 0 to 32, with larger values representing greater use severity.
Change in Specific Levels of Functioning scale (SLOF) | Baseline and 12 weeks
  An index of real-world, everyday functioning, derived by summing 30 item scores (1-5). Higher scores reflect better functioning.
Change in Behavior And Symptom Identification Scale (BASIS) - revised | Baseline and 12 weeks
  A self-report questionnaire to assess mental health treatment outcomes. Only the first 24 items (probing daily life functioning, social behavior, and mood) are included, each scored on a scale from 0 to 4. The total score is derived by summing individual item scores are re-poling some items, with larger values representing worse outcome.
Change in Serum concentrations of CBD | Baseline and 12 weeks
  To confirm bioavailability of the study drug.
Change in Serum concentrations of anandamide | Baseline and 12 weeks
  Anandamide is an endocannabinoid that has been reported to be down-regulated by cannabis use and up-regulated by CBD.

OTHER OUTCOMES:
Change in Negative Symptom Assessment (NSA-16) - exploratory | Baseline and 12 weeks
  The 16-item Negative Symptom Assessment (NSA-16) is a validated and widely used scale capturing different facets of negative symptoms. Each item is scored on a scale of 1 to 6, and the total score is derived by adding individual item scores. Larger values represent worse symptoms.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Semel Institute for Neuroscience and Human Behavior, Los Angeles, California
  - Sheppard Pratt Health System, Baltimore, Maryland
  - Maryland Psychiatric Research Center, Catonsville, Maryland

IPD SHARING:
Plan to Share IPD: No